CLINICAL TRIAL: NCT02055053
Title: A Randomized, Double-blinded, Placebo-controlled Trial of the Effects of Infusing Local Anesthesia on Post-operative Pain During Laparoscopic Inguinal Hernia Repair
Brief Title: Effects of Local Anesthesia on Post-operative Pain During Laparoscopic Inguinal Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Dmitry Nepomnayshy, Study Coordinator sub- Investigator, Lahey Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCID 2013-031
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Post Operative Pain (Post Laparoscopic Hernia Repair)
Keywords: Post Operative Pain; hernia repair
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- anesthetic intervention (Experimental): After deployment of therapeutic mesh in the preperitoneal space of the abdomen wall during the procedure, the treatment group will receive infusion of 15 cc 0.5% Bupivicaine.
  Interventions: Drug: 0.5% Bupivicaine
- Saline intervention (Placebo Comparator): After deployment of therapeutic mesh in the preperitoneal space of the abdomen wall during the procedure, the placebo group will receive the infusion of 15 cc 0.9% Saline.
  Interventions: Drug: 0.5% Bupivicaine

INTERVENTIONS:
Drug: 0.5% Bupivicaine — Local anesthetic
  Other Names: Marcaine; Sensorcaine

SUMMARY:
To assess effect of local anesthetic into the preperitoneal space during laparoscopic hernia repair on post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older with unilateral or bilateral inguinal herna for laparoscopic repair
* American Society of Anesthesiology (ASA) Class I and II

Exclusion Criteria:

* Conversion from laparoscopic to open surgery
* History of Chronic pain or ongoing treatment for chronic pain
* Age less than 18 yrs
* Allergy to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States

REFERENCES:
- [Derived] Rade M, Jayaram A, Birkett R, Ford H, Birkett D, Nepomnayshy D. A randomized, double-blinded, placebo-controlled trial of the effects of infusing local analgesia on post-operative pain during laparoscopic inguinal hernia repair. Surg Endosc. 2023 Mar;37(3):1970-1975. doi: 10.1007/s00464-022-09697-7. Epub 2022 Oct 20. PMID 36266481

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anesthetic Intervention | Saline Intervention
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anesthetic Intervention | Saline Intervention | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 35 | 35 | 70
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain Score Assessment (VAS)
Description: Pain level at 4 hours after surgery VAS scale measures pain in whole numbers from 0 (no pain) to 10 (worst imaginable pain)
Time Frame: Post-operative period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anesthetic Intervention | Saline Intervention
Number analyzed (Participants) | 35 | 35
score on a scale | 2.96 (2.3) | 3.24 (1.57)

2. Primary Outcome: Visual Analog Scale Pain Score Assessment (VAS)
Description: Pain level recorded at 3 days after surgery. VAS scale measures pain in increments of whole numbers from 0 (no pain) to 10 (most sever pain imaginable)
Time Frame: Pain scale 3 days after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anesthetic Intervention | Saline Intervention
Number analyzed (Participants) | 35 | 35
units on a scale | 3.71 (2.08) | 3.25 (1.66)

3. Secondary Outcome: Amount of Pain Medication Used in Oral Morphine Equivalents
Description: Total mg of opiate after surgery
Time Frame: 4 hours after surgery
Population: one patient's data is missing
Measure: Mean (Standard Deviation); unit: oral morphine equivalents
Arm/Group | Anesthetic Intervention | Saline Intervention
Number analyzed (Participants) | 35 | 34
oral morphine equivalents | 8.37 (12.18) | 7.72 (10.23)

4. Secondary Outcome: Duration of Narcotic Used to Control Pain
Description: Number of days post-operatively narcotic is used
Time Frame: 4 weeks post-op
Population: Data were not collected for any patients.
Arm/Group | Anesthetic Intervention | Saline Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Anesthetic Intervention | Saline Intervention
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT02055053/Prot_SAP_000.pdf